CLINICAL TRIAL: NCT06750328
Title: Procedural and Clinical Outcomes of Isolated Left Circumflex Coronary Artery Acute Occlusion in Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Outcomes of Isolated LCx Occlusion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa gamal mohammed, Resident doctor, Assiut University
Other Study IDs: LCx occlusion
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: LCx Occlusion STEMI; STEMI
Keywords: LCx occlusion STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Follow up after PPCI: To assess procedural success and short term clinical outcomes of primary PCI to isolated LCx acute

SUMMARY:
To assess procedural success and short term clinical outcomes of primary PCI to isolated LCx acute occlusion.

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) involving acute occlusion of the left circumflex (LCx) coronary artery represent only 14-21% of STEMIs

LCx acute occlusion may be difficult to be diagnosed . Only 50% of patients with LCx occlusion exhibited ST segment elevation during the acute phase, 38% showed no ST segment changes, while 15% presented with isolated ST segment depression This may lead to delay in transfer to cath lab, delay in reperfusion therapy and consequently loss of more myocytes and more major adverse cardiovascular events (MACE) .

Due to relative rare occurrence of isolated LCx coronary artery occlusion, little is known in literature about the clinical outcomes of isolated LCx occlusion , so we will conduct a retrospective observational study in our tertiary primary percutaneous coronary intervention (PCI) center to detect the incidence , procedural and clinical outcomes after 6 months of patients who had isolated LCx acute occlusion and underwent primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to Assiut University heart hospital with STEMI who underwent primary PCI that revealed isolated LCx acute occlusion (single culprit artery) between January 2018 to January 2025 will be included.

Exclusion Criteria:

-Patients with cardiogenic shock, NYHA class III-IV and multivessel coronary artery disease will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Baseline demographic, angiographic and clinical data, including cardiovascular risk factors, will be retrospectively collected. For follow up, we will contact every patient included in our study to ask about MACE.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2027-11-12 (Estimated)

PRIMARY OUTCOMES:
Complications of PPCI to LCx occlusion | 6 months
  defined as angiographic success without in-hospital complications). Angiographic success (defined as in-stent residual stenosis ≤30% without serious angiographic complications (severe coronary dissection impairing flow [type D-F], perforation, abrupt closure or no reflow) .

SECONDARY OUTCOMES:
Long follow up of outcomes of PPCI of LCx outcomes | 6 months
  The secondary endpoint will be assessment of MACE at 6 months following the index procedure. MACE ( defined as the composite of all-cause mortality, target lesion revascularization, stent thrombosis, documented atrial fibrillation and development of heart failure).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geffin R, Triska J, Najjar S, Berman J, Cruse M, Birnbaum Y. Why do we keep missing left circumflex artery myocardial infarctions? J Electrocardiol. 2024 Mar-Apr;83:4-11. doi: 10.1016/j.jelectrocard.2023.12.011. Epub 2023 Dec 26. PMID 38181483
- [Background] From AM, Best PJ, Lennon RJ, Rihal CS, Prasad A. Acute myocardial infarction due to left circumflex artery occlusion and significance of ST-segment elevation. Am J Cardiol. 2010 Oct 15;106(8):1081-5. doi: 10.1016/j.amjcard.2010.06.016. PMID 20920642
- [Background] Stribling WK, Kontos MC, Abbate A, Cooke R, Vetrovec GW, Dai D, Honeycutt E, Wang TY, Lotun K. Left circumflex occlusion in acute myocardial infarction (from the National Cardiovascular Data Registry). Am J Cardiol. 2011 Oct 1;108(7):959-63. doi: 10.1016/j.amjcard.2011.05.027. Epub 2011 Aug 4. PMID 21820644